CLINICAL TRIAL: NCT05424549
Title: A Randomized, Double-Masked, Vehicle-Controlled Crossover Clinical Trial to Assess Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of Rreproxalap in Adults With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-027
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2022-06

CONDITIONS: Dry Eye Syndromes
Keywords: dry eye disease; reproxalap; Aldeyra; ADX-102
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) dosed six times over two consecutive days
  Arms: Reproxalap Ophthalmic Solution (0.25%)
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution dosed six times over two consecutive days
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
A Randomized, Double-Masked, Vehicle-Controlled Crossover Clinical Trial to Assess Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects with Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen (18) to 70 years of age at the time of screening (either gender and any race)
2. Ability to provide written informed consent
3. Reported history of dry eye for at least 6 months prior to screening
4. Reported history of the use of eye drops for dry eye disease between 2 weeks to 6 months prior to screening

Exclusion Criteria:

1. Diagnosis of an ongoing ocular infection (bacterial, viral, or fungal), active ocular inflammation, or history of inflammatory disease (that, in the opinion of the Investigator, could interfere with study conduct or assessments) at screening
2. Contact lens use within 7 days of screening or anticipate using contact lenses during the trial
3. Systemic corticosteroid or other immunomodulatory therapy (not including inhaled corticosteroids) within 60 days of screening, or any planned immunomodulatory therapy throughout the study period
4. Women of childbearing potential (WOCBP) who are pregnant and nursing
5. If participant is of childbearing potential (female or male), unwillingness to use an acceptable means of birth control.
6. Known allergy and/or sensitivity to reproxalap or the drug product vehicle
7. A condition that the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the trial
8. Inability or unwillingness to follow instructions, including participation in all study assessments/procedures and visits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-three subjects were randomized in a crossover design.
Groups:
- Reproxalap (0.25%) First, Then Vehicle: Subjects received reproxalap six times over two consecutive days, followed by a 7-day washout, then subjects received vehicle six times over two consecutive days.
- Vehicle First, Then Reproxalap (0.25%): Subjects received vehicle six times over two consecutive days, followed by a 7-day washout, then subjects received reproxalap six times over two consecutive days.
Period: Overall Study
Arm/Group | Reproxalap (0.25%) First, Then Vehicle | Vehicle First, Then Reproxalap (0.25%)
Started | 32 | 31
Completed | 29 | 28
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproxalap (0.25%) First, Then Vehicle | Vehicle First, Then Reproxalap (0.25%) | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 59
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (13.12) | 51.2 (12.14) | 49.1 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 15 | 7 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 24 | 19 | 43
  More than one race | 0 | 5 | 5
  Unknown or Not Reported | 0 | 0 | 0
Intraocular Pressure (right eye) [Mean (Standard Deviation); unit: mmHg] | 11.6 (2.08) | 12.0 (2.76) | 11.8 (2.42)
Intraocular Pressure (left eye) [Mean (Standard Deviation); unit: mmHg] | 11.7 (1.97) | 11.6 (2.61) | 11.6 (2.29)

OUTCOME MEASURES:

1. Primary Outcome: Conjunctival Redness Assessed Via Digital Photography Over 90 Minutes in the Dry Eye Chamber
Description: Change from baseline comparison of reproxalap to vehicle for conjunctival redness assessed on a 0 to 4 scale (0 = none, 4 = extremely severe). The least squares mean (95% confidence interval) was derived from mixed model repeated measure for change from baseline included baseline as a covariate, and treatment, period, sequence, and time point as factors.
Time Frame: The efficacy assessment period was during a 90-minute dry eye chamber; baseline was pre-dose #1 for each treatment period.
Population: Intent-to-treat population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Reproxalap (0.25%): Subjects received reproxalap six times over two consecutive days.
- Vehicle: Subjects received vehicle six times over two consecutive days.
Arm/Group | Reproxalap (0.25%) | Vehicle
Number analyzed (Participants) | 61 | 61
score on a scale | 0.33 [0.23 to 0.43] | 0.44 [0.34 to 0.54]

2. Primary Outcome: Schirmer Test Mean Change From Baseline
Description: Change from baseline comparison of reproxalap to vehicle for schirmer test on a millimeter line (0 = none, 35 = maximum). The least squares mean (95% confidence interval) was derived from mixed model repeated measure for change from baseline included baseline as a covariate, and treatment, period, sequence, and time point as factors.
Time Frame: The efficacy assessment period was assessed on the first day of two consecutive dosing days for both crossover periods; baseline was pre-dose #1 for each treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Reproxalap (0.25%) | Vehicle
Number analyzed (Participants) | 61 | 61
score on a scale | -0.06 [-1.82 to 1.70] | -2.54 [-4.22 to -0.86]

ADVERSE EVENTS:
Time Frame: Two days for each intervention
Arm/Group | Reproxalap (0.25%) | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 56/61 | 2/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap (0.25%) (N=61) | Vehicle (N=60)
General disorders and administration site conditions (General disorders) | 56 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT05424549/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT05424549/SAP_001.pdf